CLINICAL TRIAL: NCT04254614
Title: A Mobile Application Guiding Patients With Inflammatory Bowel Disease During Biologic Treatment
Brief Title: Mobile Application for IBD Patients With Biologics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: NL72353.091.19
Record Dates: First submitted 2020-01-13; First posted 2020-02-05 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Biologic treatment; Mobile application
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Intervention Model Description: This is a cohort study with assessments at baseline and after implementation of the mobile application. The study period will cover 6-12 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Personalised mobile application for IBD patients (Experimental): This is a cohort study with a 1 arm intervention group, without a control group. Patients included in this study will be invited to use a mobile application. The content and functionalities of this application are described in the intervention section.
  Interventions: Device: Personalised mobile application for IBD patients

INTERVENTIONS:
Device: Personalised mobile application for IBD patients — Patients will use a mobile application for ±6months (exact period depends on interval of biologic treatment) with the following functionalities:
  * Personal interactive timeline to prepare for biologic treatment with reminders for blood tests, a questionnaire to exclude contra-indications for biologic treatment (e.g. current infection) and a message from the gastroenterology nurse when blood tests results and the questionnaire have been checked. Only in case of abnormal results or answers patients will be contacted by telephone by their gastroenterology nurse, which is currently standard care.
  * Information about the patients' diagnosis and biologic treatment.
  * General information on e.g. IBD treatment, vaccinations, frequently used medical terms, preparing for outpatient visits, what to do in case of disease symptoms.
  Patients will fill in a questionnaire to measure study outcomes at baseline and at the end of the study period.

SUMMARY:
Monitoring of biologic treatment in patients with inflammatory bowel disease (IBD) is important given the increased risk of infections. In this study we aim to evaluate the use of a mobile application to guide IBD patients and facilitate the monitoring of biologic treatment.

DETAILED DESCRIPTION:
Biologic treatment can induce and maintain remission in patients with inflammatory bowel disease (IBD). However, biologics are associated with increased risk of infections. Therefore, it is important to regularly monitor patients during the course of therapy. This process can be time consuming for patients as well as clinicians. Mobile applications, have the potential to guide patients and facilitate monitoring of biologic treatment. In this study we aim to evaluate the use of a mobile application to guide IBD patients during biologic treatment. Adult patients with diagnosis of IBD treated with biologics will be included. The mobile application with personalised content will give patients information about their treatment, reminders for example when blood tests and questionnaires to check for adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of inflammatory bowel disease
* Treatment with infliximab or vedolizumab
* Ability to read and understand Dutch language

Exclusion Criteria:

* Patients recently started with biologic treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2020-03-12 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction | 6 months
  All patients will be asked to complete questions about satisfaction with the mobile application, the information in the app and the user-friendliness of the app. This will be measured with a 7-point likert scale after using the application for ± 6 months. We will also ask patients about their overall satisfaction of care before and after implementation of the application using a visual analogue scale (VAS) scale 0 - 10.
Actual use - frequency | 6 months
  Use will be monitored with log data of the application. We will look at frequency of use of the application.
Adherence | 6 months
  The adherence of patients to reminders will be evaluated by checking time of blood tests as recorded in the electronic medical record and log data from administered questionnaires.

SECONDARY OUTCOMES:
Satisfaction of care providers | 6 months
  After ± 6 months, health care professionals will be asked to fill in a questionnaire to measure their experiences with the application, experience with monitoring the questionnaire, satisfaction, organizational advantages/disadvantages for example time investment, efficiency of work processes. This will be measured with a 7-point likert scale after using the application for ± 6 months. We will also ask care providers about their overall satisfaction with the application using a VAS scale 0 - 10.
Overall satisfaction of care providers | 6 months
  We will ask care providers about their overall satisfaction with the application using a VAS scale 0 - 10.
Number of outpatient visits | 6 months
  The total number of outpatients visits in the six months before and after implementation of the application will be compared.
Number of telephone contacts | 6 months
  The total number of telephone contacts in the six months before and after implementation of the application will be compared.
Disease and treatment knowledge | 6 months
  The knowledge of disease and its treatment of patients before and after implementation of the application will be compared and assessed using a VAS Scale (scale 0 - 10).

CONTACTS AND LOCATIONS:
Locations (1):
- Rijnstate Hospital, Arnhem, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van Erp LW, Groenen MJM, Heida W, Wisse J, Roosenboom B, Wahab PJ. Mobile application to monitor inflammatory bowel disease patients on intravenous biologic treatment: a feasibility study. Scand J Gastroenterol. 2021 Dec;56(12):1414-1421. doi: 10.1080/00365521.2021.1966832. Epub 2021 Aug 27. PMID 34448665